CLINICAL TRIAL: NCT02264587
Title: Effects and Mechanism of Mosapride Citrate on Diabetic Gastroparesis
Acronym: MDGP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liangzhou Wei (Other)
Collaborators: Sumitomo Pharma (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Liangzhou Wei, Head of departments, Qingdao University
Organization: Qingdao University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAS-IIS-2013-03
Record Dates: First submitted 2014-08-27; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Diabetic Gastroparesis
MeSH Terms: interventions — mosapride; Domperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mosapride (Experimental): mosapride 5mg by mouth, 30 minutes before meals, every times one day for 14days
  Interventions: Drug: Mosapride
- domperidone (Active Comparator): domperidone 10mg by mouth, 30 minutes before meals, every times one day for 14days
  Interventions: Drug: domperidone

INTERVENTIONS:
Drug: Mosapride — Mosapride 5mg by mouth ,3 times one day for 1 4days.
  Other Names: Gasmotin
  Arms: mosapride
Drug: domperidone — Domperidone 10mg by mouth ,3 times one day for 1 4days.
  Other Names: Motilium
  Arms: domperidone

SUMMARY:
The purpose of this study is to evaluate the effects and mechanism of mosapride citrate on diabetic gastroparesi.

DETAILED DESCRIPTION:
To evaluate the effect of mosapride on DPG by 13 C - octylic acid breath test.

IF C13- octylic acid be absorbed by mucous membrane of small intestine, octylic acid will be oxidated to CO2.Patients eating food containing C13, and then collect their expired gas at 15, 30,45,60,75,90,105,120,150,180,210,240min, analyse the mass of C13 by mass spectrometer, then can calculate the gastric emptying rate.

ELIGIBILITY:
Inclusion Criteria:

1. 18≤ age ≤ 75
2. Patients coincided to, the WHO diagnostic criteria for diabetes in 1999 (namely have diabetes symptoms, plasma glucose tendency for 11.1 / L, at any time or fasting plasma glucose tendency for 7.0 / L, or oral glucose tolerance test 2 h plasma glucose levels tendency for 11.1 / L）
3. fasting blood-glucose≤7.0mmol/L and 2h postprandial plasma glucose≤10.0mmol/L
4. Be diagnosed diabetes more than 5 years, blood sugar steady in one month.
5. have the following symptoms for over 4weeks: early satiety ,postprandial fullness ,nausea, vomting,abdominal distension,belching, inappetence, epigastric pain, constipation.
6. Be diagnosed as Delayed Gastric Emptying by C13 breath test.
7. Signed informed consent.

Exclusion Criteria:

1. take gastrointestinal drugs within 2 weeks prior to screening. Or patients with other digestive disease.
2. All patients will be administrated gastroscope in order to exclude stomach or duodenum disease, pyloric obstruction. It's normal in Liver, gallbladder, pancreas,spleen, nephridium by Ultrasound examination .
3. Serious ketoacidosis.
4. History of abdominal operation.
5. Thyroid hypofunction or hyperthyroidism.
6. nervous system disease or autoimmune diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The improvement of gastric emptying time after taking the medicine | 2 weeks
  Gastric emptying time will be tested by C13 breath test.